CLINICAL TRIAL: NCT02237859
Title: Vancomycin Prophylaxis in Recurrent Clostridium Difficile Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corewell Health West (Other)
Responsible Party: Principal Investigator, Andrew Maternowski, Physician, Corewell Health West
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 2013-303; DDI.FY14.01 (Other Grant/Funding Number: Digestive Disease Institute)
Record Dates: First submitted 2014-09-03; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Clostridium Difficile Infection
Keywords: cdiff; vancomycin; infection; clostridium difficile
MeSH Terms: conditions — Clostridium Infections; Infections | interventions — Vancomycin; Fruit and Vegetable Juices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vancomycin (Experimental): Vancomycin 125 mg PO QD vs Placebo
  Interventions: Drug: Vancomycin; Dietary Supplement: fruit juice/placebo

INTERVENTIONS:
Drug: Vancomycin — Vancomycin Group: Study participants started on a broad-spectrum antibiotic will be initiated on Vancomycin 125 mg PO QD within 48 hrs of the 1st dose of primary broad-spectrum antibiotic and continued to complete a 10 day course regardless of the duration of primary antibiotic. Dose of oral Vancomycin is 125 mg PO QD. Vancomycin liquid will be dissolved in fruit juice which is standard practice at Spectrum Health Hospitals. Both groups will continue in the study even if their broad spectrum antibiotic therapy is curtailed prior to 10 days.
Dietary Supplement: fruit juice/placebo — Placebo Group: Will receive similar volume of fruit juice/placebo for 10 days.

SUMMARY:
We are doing this research study to determine if taking vancomycin in addition to a broad-spectrum antibiotic will decrease the chance of developing recurrent Clostridium difficile infection.

DETAILED DESCRIPTION:
To determine whether prophylactic use of oral vancomycin reduces the incidence of recurrent Clostridium difficile infection (RCDI) in hospitalized patients admitted from their home or another health care facility (HCF) who are exposed to concurrent broad spectrum antibiotics.

This is a randomized research study, which means that the treatment you get will be chosen by chance, like flipping a coin. You will have a 50/50 chance of receiving one of the following:

1. Group 1 (Treatment Group): single daily dose of vancomycin in liquid form (study medication).
2. Group 2 (Placebo Group): single daily dose of placebo (a placebo will look just like the study medication, but contains no medication, only a substance like sterile water).

Depending on the group you are placed in (which is chosen by a computer), you will receive either a daily dose of the study medication or a daily dose of the placebo for a total of ten days. If you are discharged from the hospital prior to ten days, you will be given the study medication to complete outside of the hospital with written instructions.

A member of the Research staff will monitor you daily during the 10 days of treatment for any adverse reactions or any signs and symptoms of recurrent Clostridium difficile infection. If you are discharged prior to ten days, the monitoring will take place via telephone call daily until completion of the ten day treatment.

You will be contacted again by telephone at 1, 3, and 6 months after completion of the study medication to inquire about your general health and any changes in health status.

Other medical information from your records and charts may also be collected by us for purposes of review for this study.

ELIGIBILITY:
Inclusion Criteria:

1. In patients >19 years of age
2. History of C. difficile diarrhea within 16 weeks and treated with Flagyl or Vancomycin during last episode.
3. Patients started on antibiotics during current admission for any other indication at any point of time during hospital course.

Exclusion Criteria:

1. Current diagnosis of CDI
2. First episode of CDI during this admission.
3. Allergy to Vancomycin or other known intolerance
4. Pregnant

h) Patient has received broad-spectrum antibiotics for more than 48 hours for this admission j) Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of recurrent Clostridium difficile infection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Maternowski, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health Hospital, Grand Rapids, Michigan, United States